CLINICAL TRIAL: NCT02795013
Title: Genetic Study of Families With High Frequency of Hodgkin Lymphoma
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: HudsonAlpha Institute for Biotechnology (Other)
Responsible Party: Sponsor
Other Study IDs: FAMHL
Record Dates: First submitted 2016-06-06; First posted 2016-06-09 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Hodgkin Lymphoma
Keywords: Genetic studies; Pediatric
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva, minimal blood, or tumor will be retained for whole exome sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with Hodgkin Lymphoma: Those with a confirmed diagnosis of Hodgkin Lymphoma (HL) and family members who consent and enroll in this study.
- Family Members without Hodgkin Lymphoma: Those unaffected by HL will serve as a control group to compare with those with HL.

SUMMARY:
Hodgkin lymphoma (HL) is a relatively rare disorder with known familiar aggregation (i.e. HL in more than one child, or parent and child). Because affected individuals in familial HL are genetically related, the existence of such families has long been considered as evidence in support of a genetic basis of HL susceptibility. However, it is largely unknown which genetic variations are responsible for recurring HL in families. Because the effects of genetic variants are likely to be strong in familial HL, identification of such variations will potentially reveal biological pathways critical to the pathogenesis of HL.

PRIMARY OBJECTIVE:

* To perform genome-wide sequencing of families with recurring Hodgkin lymphoma cases (affected as well as non-affected family members) to identify potential disease-causing germline genetic variations.

SECONDARY OBJECTIVE:

* To describe demographic and clinical features of the affected families.

DETAILED DESCRIPTION:
This study entails a clinical interview and submission of a peripheral blood or saliva sample for non-tumor DNA. Participants diagnosed with HL at outside institutions will be requested to sign a release form to allow the outside institution to send their pathology report confirming their HL diagnosis. If available, previously banked tumor tissue samples will be utilized to assess genetic alterations related to HL. Detailed history will be obtained (e.g., demographics, environmental exposures, cancer risk factors, and family pedigree) to facilitate the analysis of phenotype-genotype correlations, taking into account potential confounding factors.

Investigators will examine the germline and possibly the tumor DNA of each individual participant and use the data from all participants to determine if a gene change is related to HL.

ELIGIBILITY:
Inclusion Criteria:

* Patient with HL diagnosed ≤ 21 years of age with a first-degree relative also diagnosed with HL.
* Family members of the patient, either affected or unaffected by a malignancy who agree to participate in the study.
* Research participant or legal guardian, as appropriate, must provide informed consent for this protocol.

Exclusion Criteria:

* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of Hodgkin Lymphoma (HL), and family members of the patient, either affected or unaffected by a malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Germline genetic variations | Once, within 1 month of enrollment
  Whole exome sequencing of affected and unaffected individuals in these families will be performed. Genetic variants potentially related to HL will be identified on the basis of its co-segregation with HL disease status (e.g., unique variants in individuals affected by HL would be considered as risk variants). Family members without HL (regardless of any other history of malignancy) will be considered as control and be compared against members with HL.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Flerlage, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols